CLINICAL TRIAL: NCT00007059
Title: Study of the Pharmacokinetics of Mycophenolate Mofetil in Patients Who Have Undergone Orthotopic Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of North Carolina (Other)
Purpose: Treatment
Other Study IDs: NCRR-M01RR00046-1404; UNCCH-GCRC-1404; ROCHE-CEL028
Record Dates: First submitted 2000-12-06; First posted 2000-12-07 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Graft Versus Host Disease
Keywords: disease-related problem/condition; graft versus host disease; rare disease
MeSH Terms: conditions — Graft vs Host Disease; Rare Diseases | interventions — Mycophenolic Acid

INTERVENTIONS:
Drug: mycophenolate mofetil

SUMMARY:
OBJECTIVES: I. Determine the effects of bile externalization and antibiotic gut sterilization on the pharmacokinetics of mycophenolate mofetil in patients who have undergone orthotopic liver transplantation.

II. Correlate serum concentrations of mycophenolic acid with inosine monophosphate dehydrogenase activity in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients begin a mycophenolate mofetil (MMF)-containing regimen within the first 5 days after transplantation. Patients have blood drawn on postoperative days 7, 21, 42, 70, 98, 126, and 154. Urine is collected on postoperative days 7, 21, and 42. Patients with T-tube bile externalization also have bile collected on postoperative day 7.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

Orthotopic liver or kidney transplant recipients who started on a mycophenolate mofetil-containing immunosuppressive regimen within 5 days after transplant

Kidney transplant recipients will serve as study controls

--Prior/Concurrent Therapy--

* No concurrent bile acid sequestrants
* No mycophenolate mofetil as part of rescue therapy regimen
* No concurrent albumin replacement therapy

--Patient Characteristics--

Renal: Urine output at least 500 mL/day OR Creatinine less than 2.5 mg/dL

Other:

* Not pregnant
* No mental incompetency
* No prisoners or parolees HIV negative
* No active infection defined as: Temperature above 101 F with WBC greater than 12,000/mm3 and left shift OR Two or more positive cultures of a single isolated organism from blood, urine, or sputum

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 1998-06

CONTACTS AND LOCATIONS:
Overall Officials: Robert E. Dupuis, Study Chair — University of North Carolina
Locations (1):
- University of North Carolina School of Medicine, Chapel Hill, North Carolina, United States